CLINICAL TRIAL: NCT01310842
Title: Social Determinants and Smoking Cessation
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010-0950; RP110025 (Other Grant/Funding Number: CPRIT); 1K99MD010468-01 (NIH)
Record Dates: First submitted 2011-02-21; First posted 2011-03-09 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation
Keywords: Smoker; Smoking Cessation; Social Determinants; Environmental Effects; Individual-level effects; Nicotine patch; Smart Phone; SP; Global Positioning System; GPS; Questionnaires; Saliva samples
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples at Baseline, week 12, and week 26 visits collected for cotinine tests.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pilot Smoking Cessation: 4 weeks nicotine patch therapy, self-help materials, and 5 in-person counseling sessions.
  Interventions: Behavioral: Questionnaires; Drug: Nicotine Patch Therapy; Behavioral: Counseling Sessions
- Smoking Cessation: 4 weeks nicotine patch therapy, self-help materials, and 7 in-person counseling sessions.
  Interventions: Behavioral: Questionnaires; Drug: Nicotine Patch Therapy; Behavioral: Counseling Sessions

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed at each study visit, taking 60-90 minutes, in addition to 4 Smart Phone initiated assessments per day during waking hours, taking about 5-10 minutes.
  Other Names: Survey
Drug: Nicotine Patch Therapy — 4 weeks of nicotine patch therapy
Behavioral: Counseling Sessions — 5 or 7 in person counseling sessions on smoking cessation: Baseline, Week 0/Quit Date (1 week following the baseline visit), Week 1, Week 2, Week 3 for Pilot Group and additional sessions Week 12 and Week 26 for other group.

SUMMARY:
The goal of this study is to learn about the influence of the social and physical environment on smoking cessation (quitting smoking) among smokers.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will receive help to quit smoking, including written self-help materials, counseling, and a supply of the nicotine patch. Over the next 6 months, you will visit MD Anderson 7 times.

Study Visits:

Your first visit is the "baseline" visit when you enter the study. You will then attend 6 additional in-person visits: Week 0 (1 week after the baseline visit), Week 1, Week 2, Week 3, Week 12, and Week 26.

During the baseline visit you will receive a small, hand-held personal phone and be trained in how to use it. You will carry this phone with you for 4 weeks. You will use the phone to answer questions about your mood, stress, and smoking-related issues. You will be asked to fill out some questions on the phone each time you have an urge to smoke. Also, the phone will "beep" at random and set times and ask that you answer some questions. This phone will not wake you during the night and you will be able to wait to answer questions for a few minutes if it goes off when you are busy. Answering the questions should take about 5-10 minutes. This small, hand-held personal phone will also have a GPS system activated that will record where you are during the waking hours every day while you are on study.

Study Tests:

The following tests and procedures will be performed at each study visit:

* You will complete some questionnaires that will include questions about your feelings, moods, and smoking status. These will take 60-90 minutes to complete.
* You will complete a breath test to help estimate (guess) the amount of cigarette smoke you inhale. The breath test uses a disposable cardboard tube that is attached to the machine, and you blow a long, slow, steady breath into it.
* At the baseline, Week 12, and Week 26 visits, you will have saliva samples collected for cotinine tests. To collect the saliva, you will be asked to put a small piece of cotton in your mouth for a few minutes. These samples will be used to measure the amount of cotinine in your saliva. Cotinine is a chemical released in your body when it breaks down nicotine.
* You will have your height, weight, and waistline measured.

You may be contacted by mail, telephone, and/or e-mail during the study to be given reminders of clinic visits. You will be asked to provide the names and contact information for family and/or friends for the study staff to contact if the study staff has trouble reaching you.

Length of Study:

You will be considered off study when you complete the Week 26 visit.

After you return the phone and GPS, all of your information that is stored on the devices will be erased. After the information is erased from the devices, it cannot be retrieved.

This is an investigational study. The nicotine patch used in this study is FDA approved and commercially available. You will receive 4 weeks of nicotine patches.

Up to 300 smokers will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 and above
2. Current smoker with a history of at least 5 cigarettes/day for the last year (participant must register a CO level of 8 or higher)
3. Motivated to quit within the next 30 days
4. Valid home address reflective of residence in Houston
5. Functioning telephone number
6. Can speak, read, and write in English
7. Marginal or adequate health literacy

Exclusion Criteria:

1. Contraindication for nicotine patch use
2. Regular use of tobacco products other than cigarettes (cigars, pipes, smokeless tobacco)
3. Use of nicotine replacement therapy products or other smoking cessation medications, other than the nicotine patches supplied during the study
4. Pregnancy or lactation
5. Another household member is enrolled in this protocol
6. Active substance abuse problem
7. Scores below the 6th grade literacy level on the Rapid Estimate of Adult Literacy in Medicine (REALM)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current smoker, age 18 years or above, with a history of at least 5 cigarettes/day for the last year and resides in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Influence of Social and Physical Environment on Smoking Cessation Among Smokers | 3 weeks
  Participants followed from 2 weeks prior to quit date through 26 weeks after quit date, assessed for 4 contiguous weeks (1 week precessation through 3 weeks postcessation) using state-of-the-science ecological momentary assessment (EMA) and global positioning system (GPS) procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin L. Strong, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org